CLINICAL TRIAL: NCT03037814
Title: Clinical Performance of Restorative Materials in Class II Cavities of Primary Molar Teeth
Brief Title: Clinical Performance of Restorative Materials in Primary Teeth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zafer Cavit Cehreli, DDS, PhD, Prof, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUDHF-3-primary teeth
Record Dates: First submitted 2017-01-29; First posted 2017-01-31 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Caries; Dentin; Dental Caries
Keywords: restorative materials; primary teeth; children
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Compomer (Other): Adhesive agent+Compomer
  Interventions: Device: RMGIC; Device: Giomer; Device: Amalgam
- RMGIC (Other): Primer+RMGIC
  Interventions: Device: Compomer; Device: Giomer; Device: Amalgam
- Giomer (Other): Adhesive Agent+ Giomer
  Interventions: Device: Compomer; Device: RMGIC; Device: Amalgam
- Amalgam (Other): Amalgam
  Interventions: Device: Compomer; Device: RMGIC; Device: Giomer

INTERVENTIONS:
Device: Compomer — Aesthetic resin dental materials that are used to replace structure loss, commonly for dental caries of primary tooth. Compomers designed to combine the aesthetics of traditional composite resins with the fluoride release and adhesion of glass-ionomer cements.
  Arms: Amalgam; Giomer; RMGIC
Device: RMGIC — Dental restorative materials that are a combination of the desirable properties of glass-ionomer (fluoride release and chemical adhesion) with high strength and low solubility of resins.
  Arms: Amalgam; Compomer; Giomer
Device: Giomer — Giomers are dental materials that are hybrid of compomers and glass ionomers, and are used to restore dental caries.
  Arms: Amalgam; Compomer; RMGIC
Device: Amalgam — Amalgam is a silver-colored dental restorative material that can be used to restore both primary and permanent posterior teeth which have dental caries.
  Arms: Compomer; Giomer; RMGIC

SUMMARY:
The purpose of this study is to evaluate and compare the clinical performance of dental restorative materials in Class II cavities of primary molar teeth

DETAILED DESCRIPTION:
Restorations will be placed on four primary molar teeth with proximal caries, in a split mouth design. 100 patients will be included in the study. The teeth will be randomized into four groups according to the restorative materials.

Group 1: Adhesive agent+ Compomer (Dyract AP, Dentsply DeTrey, Konstanz,Germany) Group 2: Primer + Resin modified glass ionomer (Vitremer, 3M ESPE, U.S.) Group 3: Adhesive agent + Giomer (Beautifil II, (Shofu Dental, Tokyo, Japan) Group 4: Amalgam (Permite amalgam, SDI Limited, Bayswater, Australia) The restorations will be evaluated at baseline, 3., 6., 12. months for the first year, and at every 6 months for 5 years. The modified US Public Health Service criteria (secondary caries, marginal integrity, marginal discoloration and retention) will be used for clinical evaluation of restorations. The data will be analysed statistically using Wilcoxon test, chi square test and the Kaplan-Meier survival method will be used to estimate survival percentages.

ELIGIBILITY:
Inclusion Criteria:

* Patients and parent of the patients who accept to participate and sign the informed consent
* Patients who have at least four first and/or second primary molars with proximal caries that require class II restorations
* Teeth that have healthy lamina dura and periodontal ligament
* Teeth that have caries lesions extending no more than the outher half of dentin radiographically

Exclusion Criteria:

* Patients and parent of the patients who don't accept to participate and sign the informed consent
* Teeth that are previously restored
* Patients who are uncooperative
* Teeth that doesn't have proximal or occlusal contacts with adjacent healthy teeth
* Patients who have bruxism, skeletal or dental malocclusion
* Teeth that have developmental defects or anomalies

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-09-28 (Estimated); Primary Completion 2026-07-25 (Estimated); Study Completion 2027-03-25 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of restorative materials in class II cavities on primary molar teeth according to the modified USPHS criteria | 5 years
  Long-term clinical success of different restorative materials in class II cavities on primary molar teeth

CONTACTS AND LOCATIONS:
Overall Officials: Zafer C Cehreli, DDS, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Clinical Study Report: 26161601 — http://www.ncbi.nlm.nih.gov/pubmed/26161601
- Available data/document: Clinical Study Report: 19953810 — http://www.ncbi.nlm.nih.gov/pubmed/19953810
- Available data/document: Clinical Study Report: 12542617 — http://www.ncbi.nlm.nih.gov/pubmed/12542617